CLINICAL TRIAL: NCT02997436
Title: Asa Test ; un Nouvel Outil Dans le dépistage du Traitement Par Aspirine ? (This Official Titre is in French and Contains no Spelling Error. English Translation for it Would be : "ASA-test. A New Tool for the Screening of Aspirin Treatment")
Brief Title: First Approach for Aspirin Misuse Objective Screening
Acronym: FirstAMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01157-44
Record Dates: First submitted 2016-12-06; First posted 2016-12-20 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2016-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PAD patients (Experimental): Patients referred for vascular ultrasound investigation for suspicion of peripheral artery disease (PAD).
  Intervention is measurement of microvascular response to current application on the skin by Laser speckle flowmetry
  Interventions: Device: Laser speckle flowmetry

INTERVENTIONS:
Device: Laser speckle flowmetry — A galvanic current (0.1 mA) will be applied between 2 patches on the forearm of patient and protocol was repeated at 4 minutes.
  Microvascular response to current application (CIV) will be recorded by laser speckle flowmetry 10 minutes later.
  Measurement of the value of skin blood flow (by laser speckle) at the stimulated area as compare to a non stimulated adjacent skin value taken as a reference Usual treatment will be recorded

SUMMARY:
prospective interventional study. The aim is to analyse the effect of usual ongoing treatments over the microvascular cutaneous response to galvanic current application (Current induced vasodilation ; CIV) on the forearm of subjects referred for ultrasound investigations due to suspicion of peripheral artery disease. Hypothesis is that the use of aspirin (even at low dose) abolishes the response .

DETAILED DESCRIPTION:
At admission eligible patients are proposed to participate. Written consent is signed after complete oral and written explanation of the protocol is signed.

No register of non-included patients will be kept. In included patients, in parallel to the routine ultrasound investigation for which the patient is referred, microvascular investigation will be performed as explained later in arm description.

Usual ongoing treatments are obtained by history and recorded. The end of the visit is the end of the participation of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* subjects referred for investigation of peripheral arterial disease.
* Affiliation to the French National healthcare system
* French speaking patients
* Ability to stand still for half a minute.

Exclusion Criteria:

* pregnancy
* inability to understand the study goal
* Patients protected by decision of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
correlation of treatments to CIV response. | 10 minutes after the second period of current application
  Classification of drugs in drug type categories. encoding in 1 (presence) or 0 ug (absence) of the drug category in the usual treatment of the patient. Multiple regression analysis of the different drug categories as factors influencing the increase in skin blood flow after CIV.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Sophie Fernandez, MD, Principal Investigator — UH Angers; Pierre Abraham, MD, PhD, Principal Investigator — UH Angers; Philippe Bouye, MD, Principal Investigator — UH Angers; Valmont Richard, MD, Principal Investigator — UH Angers; Vincent Azzola, MD, Principal Investigator — UH Angers
Locations (1):
- UH Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No